CLINICAL TRIAL: NCT04738942
Title: An Open-Label, Phase 3 Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Intravenous (IV) Vedolizumab Administered Every 4 Weeks (Q4W) in Japanese Patients With Moderate to Severe Ulcerative Colitis or Crohn's Disease Who Experienced Secondary Loss of Response During Maintenance Therapy With Vedolizumab IV Administered Every 8 Weeks (Q8W)
Brief Title: A Study of Intravenous Vedolizumab Administered Every 4 Weeks in Japanese Participants With Moderate to Severe Ulcerative Colitis or Crohn's Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-3039; U1111-1262-7325 (Other: WHO); jRCT2031200371 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vedolizumab 300 mg in UC cohort (Experimental): Vedolizumab 300 mg, IV infusion, for up to 12 weeks Q4W for Treatment phase, and until the date of marketing approval of vedolizumab IV Q4W or study termination for Extension phase.
  Interventions: Drug: Vedolizumab
- Vedolizumab 300 mg in CD cohort (Experimental): Vedolizumab 300 mg, IV infusion, for up to 12 weeks Q4W for Treatment phase, and until the date of marketing approval of vedolizumab IV Q4W or study termination for Extension phase.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab 300 mg, IV infusion

SUMMARY:
The main aim of the study is to learn if 4-weekly vedolizumab improves symptoms of Japanese participants with moderate to severe ulcerative colitis (UC) or Crohn's disease (CD). Vedolizumab is commercially available in Japan for 8-weekly treatment but not for 4-weekly treatment.

The study doctors will also monitor side effects from the study treatment.

This study will take place in Japan.

At the first visit, the study doctor will check if each person can take part. For those who can take part, participants will receive vedolizumab intravenously once every 4 weeks. After 3 infusions of vedolizumab (which will be 12 weeks of treatment), the study doctor will assess if symptoms of the participants have improved.

Participants who do not have improved symptoms after 12 weeks of treatment with vedolizumab will stop this treatment. Then, they will visit the study clinic 16 weeks after their last infusion of vedolizumab for a final check-up.

Participants who have improved symptoms after 12 weeks of treatment with vedolizumab will continue to receive vedolizumab every 4 weeks. Then, after their last infusion of vedolizumab, the participants will visit the study clinic 16 weeks later for a final check-up. Finally, the study clinic will make a phone call to each participant 6 months after their last infusion to check if they have any health problems.

ELIGIBILITY:
Inclusion Criteria:

UC cohort

1. The participant has moderate to severe UC, who had previously shown clinical response in initial treatment with commercially available vedolizumab IV, then experienced secondary loss of response during maintenance therapy with commercially available vedolizumab IV Q8W.

   Previous "clinical response" is to be judged by the investigators referring to one of the following criteria.
   * Reduction of >=2 points and >=25% in modified Mayo score, and a decrease of >=1 point in rectal bleeding subscore or rectal bleeding subscore of =<1, from the start of initial treatment with commercially available vedolizumab IV.
   * Reduction of >=2 points and >=25% in partial Mayo score, and a decrease of >=1 point in rectal bleeding subscore or rectal bleeding subscore of =<1, from the start of initial treatment with commercially available vedolizumab IV.
   * Significant improvement on endoscopy (i.e., a decrease of >=2 points in Mayo endoscopic subscore).

   "Secondary loss of response" is to be judged by the investigators referring to one of the following criteria.
   * Increase of >=2 points in modified Mayo score, and an increase of >=1 point in rectal bleeding subscore or rectal bleeding subscore >=2, from the start of maintenance therapy with commercially available vedolizumab IV.
   * Increase of >=2 points in partial Mayo score, and an increase of >=1 point in rectal bleeding subscore or rectal bleeding subscore >=2, from the start of maintenance therapy with commercially available vedolizumab IV.
   * Significant deterioration on endoscopy (i.e., an increase of >=2 points in Mayo endoscopic subscore).
2. The participant has active UC as determined by a modified Mayo score of >=5 at baseline (within 10 days prior to the start of treatment phase), with a Mayo rectal bleeding subscore of >=1 at baseline (within 10 days prior to the start of treatment phase) and a Mayo endoscopic subscore of >=1 as assessed by the central reader.

CD cohort

1. The participant has moderate to severe CD, who had previously shown clinical response in initial treatment with commercially available vedolizumab IV, then experienced secondary loss of response during maintenance therapy with commercially available vedolizumab IV Q8W.

   Previous "clinical response" is to be judged by the investigators referring to one of the following criteria.
   * Reduction of >=70 points in CDAI score from the start of initial treatment with commercially available vedolizumab IV.
   * Reduction of >=3 points in HBI score from the start of initial treatment with commercially available vedolizumab IV.

   "Secondary loss of response" is to be judged by the investigators referring to one of the following criteria.
   * Increase of >=70 points in CDAI score from the start of maintenance therapy with commercially available vedolizumab IV.
   * Increase of >=3 points in HBI score from the start of maintenance therapy with commercially available vedolizumab IV.
2. The participant has active CD as determined by a CDAI score of >=220 at baseline (within 10 days prior to the start of treatment phase).
3. The participant has a C-reactive protein (CRP) level >3.0 mg/L during the screening phase.

Exclusion Criteria:

1. The participant has had extensive colonic resection, subtotal or total colectomy.
2. The participant has received any of the investigational or approved non-biologic therapies (e.g., cyclosporine, tacrolimus or tofacitinib, except for those specifically listed as permitted medications) for the treatment of underlying disease within 30 days or 5 half-lives of screening (whichever is longer).
3. The participant has received any investigational or approved biologic or biosimilar agent other than vedolizumab within 60 days or 5 half-lives of screening (whichever is longer).
4. The participant has a clinically significant active infection (e.g., pneumonia, pyelonephritis or coronavirus disease 2019 [COVID-19]) within 30 days prior to screening or during screening, or has an ongoing chronic infection.
5. The participant has known or suspected intolerance or hypersensitivity to vedolizumab or closely related compounds, or any of the vedolizumab IV excipients.
6. The participant has active cerebral/meningeal disease, or signs/symptoms of progressive multifocal leukoencephalopathy (PML) or any history of PML at screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Response at Week 12 Based on Modified Mayo Score in UC Cohort | Week 12
  Clinical response is defined as a reduction of >=2 points and >=25% in modified Mayo score, and a decrease of >=1 point in rectal bleeding subscore or rectal bleeding subscore of =<1 from baseline (Week 0). Mayo score is an instrument designed to measure disease activity of UC. Modified Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and Mayo endoscopic subscore (findings on endoscopy), each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher score indicates more severe disease.
Percentage of Participants with Clinical Response at Week 12 in CD Cohort | Week 12
  Clinical response is defined as a reduction of =>70 points in CDAI score from baseline (Week 0). CDAI assesses CD based on clinical signs and symptoms such as number of liquid stools, intensity of abdominal pain, general well being, presence of comorbid conditions, use of antidiarrheal, physical examination and laboratory findings. Total score ranges from 0 to 600 points. Higher score indicates more severe disease.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 12 Based on Modified Mayo Score in UC Cohort | Week 12
  Clinical remission is defined as a modified Mayo score of =<2, and no individual subscore >1. Mayo score is an instrument designed to measure disease activity of UC. Modified Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and Mayo endoscopic subscore (findings on endoscopy), each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher score indicates more severe disease.
Percentage of Participants with Mucosal Healing at Week 12 in UC Cohort | Week 12
  Mucosal healing is defined as a Mayo endoscopic subscore of =<1, in participants with baseline Mayo endoscopic subscore of >=2. Mayo score is an instrument designed to measure disease activity of UC.
Percentage of Participants with Corticosteroid-Free Remission Based on Partial Mayo Score in UC Cohort | Week 12
  Corticosteroid-free remission is defined as participants using oral corticosteroids at baseline (Week 0) who have discontinued oral corticosteroids and are in clinical remission based on partial Mayo score at Week 52. Clinical remission based on partial Mayo score is defined as a partial Mayo score of =<2, and no individual subscore >1. Mayo score is an instrument designed to measure disease activity of UC. Partial Mayo score consists of 3 sub-scores: stool frequency, rectal bleeding, and physician's global assessment, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher scores indicates more severe disease.
Percentage of Participants with Clinical Remission at Week 12 in CD Cohort | Week 12
  Clinical remission is defined as a CDAI score of =<150. CDAI assesses CD based on clinical signs and symptoms such as number of liquid stools, intensity of abdominal pain, general well being, presence of comorbid conditions, use of antidiarrheal, physical examination and laboratory findings. Total score ranges from 0 to 600 points. Higher score indicates more severe disease.
Percentage of Participants with Enhanced Clinical Response at Week 12 in CD Cohort | Week 12
  Enhanced clinical response is defined as a reduction of >=100 points in CDAI score from baseline (Week 0). CDAI assesses CD based on clinical signs and symptoms such as number of liquid stools, intensity of abdominal pain, general well being, presence of comorbid conditions, use of antidiarrheal, physical examination and laboratory findings. Total score ranges from 0 to 600 points. Higher score indicates more severe disease.
Percentage of Participants with Corticosteroid-Free Remission in CD Cohort | Week 12
  Corticosteroid-free remission is defined as participants using oral corticosteroids at baseline (Week 0) who have discontinued oral corticosteroids and are in clinical remission at Week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (20):
- Japan (20):
  - Ieda Hospital, Toyota, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Tsujinaka Hospital, Kashiwa, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Sapporo Kosei General Hospital, Sapporo, Hokkaido
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - Ofuna Chuo Hospital, Kamakura, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Institute of Science Tokyo Hospital, Bunkyo-ku, Tokyo
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Infusion Clinic., Osaka
  - Osaka Metropolitan University Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/6037f111e732fe001e0b88fd